CLINICAL TRIAL: NCT07275008
Title: Efficacy and Long-term Prognosis of Auxiliary Liver Transplantation
Brief Title: Efficacy and Prognosis of Auxiliary Liver Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Zhi-Jun Zhu (Other)
Responsible Party: Sponsor-Investigator, Zhi-Jun Zhu, Professor, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: BFH20251127004
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Liver Transplantation; Auxiliary Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected at 3 days, 7 days, 14 days, 1 month, and 3 months postoperatively for Olink proteomics analysis. Peripheral blood mononuclear cells (PBMCs) were isolated for flow cytometry detection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- auxiliary liver transplantation: Patients who underwent auxiliary liver transplantation at our center during the study period
- living donor liver transplantation: Patients who underwent traditional orthotopic living donor liver transplantation at our center during the study period.

SUMMARY:
The objective of this observational study is to systematically compare the efficacy and patient prognosis between auxiliary liver transplantation and living donor liver transplantation, and to explore the postoperative recovery, survival rate, rejection, postoperative complications, and long-term prognosis of patients undergoing auxiliary liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent auxiliary liver transplantation or living donor liver transplantation (LDLT).
2. Patients with complete medical records and follow-up data.

Exclusion Criteria:

1. Patients who underwent retransplantation.
2. Patients who underwent other organ transplantation (or multiorgan transplantation).
3. Patients with severe missing postoperative follow-up data or loss to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were treated at the Liver Transplantation Center of Beijing Friendship Hospital, Capital Medical University between December 2025 and December 2028, and who underwent either auxiliary liver transplantation (study group) or conventional liver transplantation (control group).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Within one year after liver transplantation

SECONDARY OUTCOMES:
Complications | Within one year after liver transplantation
  Rejection, vascular, biliary and other related complications
changes in peripheral blood lymphocytes | within 3 months after liver transplantation
  Peripheral blood lymphocytes during the early post-transplant period were compared between the auxiliary and living donor liver transplantation groups to identify differences.

IPD SHARING:
Plan to Share IPD: No